CLINICAL TRIAL: NCT02002897
Title: Fractional Carbon Dioxide Laser Versus UVA1 Phototherapy for Treatment of Localized Scleroderma: A Clinical & Immunohistochemical Comparative Study
Brief Title: Fractional Carbon Dioxide Laser Versus UVA 1 in Treatment of Localized Scleroderma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzan Shalaby, Assisstant lecturer - Dermatology department - Faculty of medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDCU-24684
Record Dates: First submitted 2013-09-05; First posted 2013-12-06 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Localized Scleroderma
Keywords: Localized scleroderma UVA1 fractional carbon dioxide laser
MeSH Terms: conditions — Scleroderma, Localized

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fractional carbon dioxide laser (Experimental): Single session of fractional laser is done using DEKA machine , for 3 months .
  Interventions: Device: Fractional carbon dioxide laser
- Ultraviolet A1 phototherapy (UVA1) (Active Comparator): 24 sessions of UVA 1 phototherapy are give at a rate of 3 sessions per week , at a dose of 30 joules using a Waldman targeted machine.
  Interventions: Device: Ultraviolet A1 phototherapy (UVA1)

INTERVENTIONS:
Device: Fractional carbon dioxide laser — Fractional carbon dioxide laser (10,600 nm), a session once per month, total of 3 sessions with full clinical evaluation and investigations before and one month after the last session of treatment.
  Arms: Fractional carbon dioxide laser
Device: Ultraviolet A1 phototherapy (UVA1) — localized UVA1 phototherapy (340-400 nm), low dose irradiation, at a rate of 3 sessions per week , total of 24 sessions with full clinical evaluation and investigations before and after treatment and clinical follow up one month after treatment.
  Arms: Ultraviolet A1 phototherapy (UVA1)

SUMMARY:
The study aims at evaluating the efficacy of the fractional carbon dioxide laser as a new modality for treatment of localized scleroderma and to compare its results with the well established method of UVA 1 phototherapy.

DETAILED DESCRIPTION:
The study includes 20 Cases presenting with one or more lesions of morphea (plaque, linear and atrophic). Each case will be subjected to:

1. -Informed consent. 2-Detailed history 3- Clinical examination to assess type, site, extent. 4-Clinical evaluation before treatment, in the follow up period and after treatment ( 24 sessions of UVA1) (one month after last CO2 laser session) using a scoring system:

   * Skin thickness: 0-3, 0: normal; 1: thickened skin; 2: decreased ability to move the skin; 3: unable to pinch or move skin (according to the Modified Rodnan skin score)
   * Dermal atrophy: 0-3, 0: none, 1: shiny, 2: visible vessels, 3: obvious atrophy
   * Dyspigmentation (Hypo or hyper pigmentation): 0-3, 0: none, 1: mild, 2: moderate ,3: marked C- Digital Photography before, follow up and after treatment using the same digital camera , at fixed distance and constant settings for standardization .

     5-Investigations: A- Punch biopsy: A punch biopsy will be taken before and after treatment to be stained with haematoxylin and eosin.

B-Immunohistochemical assessment of

* MMP1 (matrix metalloproteinase 1) in the pre and post treatment skin biopsies.
* TGFß ( transforming growth factor beta)in the pre and post treatment skin biopsies.

  6-Treatment intervention: Two lesions with identical scoring will be chosen for the treatment interventions.
  1. Lesion number (1) will be subjected to: localized UVA1 phototherapy (340-400 nm), low dose irradiation, at a rate of 3 sessions per week , total of 24 sessions with full clinical evaluation and investigations before and after treatment and clinical follow up one month after treatment.
  2. Lesion number (2) will be subjected to: Fractional carbon dioxide laser (10,600 nm), a session once per month, total of 3 sessions with full clinical evaluation and investigations before and one month after the last session of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Types of morphea: plaque, linear and atrophic.
2. Patients are either new or discontinued systemic treatment for at least two months

Exclusion Criteria:

1. Morphea profunda and systemic scleroderma (diagnosed by: Rayaund's Phenomenon and sclerodactyly +/- internal organ affection)
2. Contraindications to phototherapy: eg: photosensitivity, systemic lupus, melanoma, skin cancer, or porphyria.
3. Contraindications to laser: Use of systemic retinoids in the last 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of fractional carbon dioxide laser as a new method for treatment of localized scleroderma | 4 months
  Efficacy will be evaluated by clinical assessment by blinded physician , biopsy before and after treatment for collagen assessment , Ultrasound bio-microscopy before and after treatment and patient satisfaction scores .

SECONDARY OUTCOMES:
Assessing the degree of improvement of cases of localized scleroderma using each method | 4 months
  Improvement will be evaluated by clinical assessment by blinded physician , biopsy before and after treatment for collagen assessment , Ultrasound bio-microscopy before and after treatment and patient satisfaction scores .

OTHER OUTCOMES:
Assessing the complications of each type of therapy | 4 months
  check list for each of common complications of Laser therapy & photo therapy is done for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan M Shalaby, Ass.lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University- Dermatology outpatient clinic, Cairo, Egypt

REFERENCES:
- [Background] Kineston D, Kwan JM, Uebelhoer NS, Shumaker PR. Use of a fractional ablative 10.6-mum carbon dioxide laser in the treatment of a morphea-related contracture. Arch Dermatol. 2011 Oct;147(10):1148-50. doi: 10.1001/archdermatol.2011.247. No abstract available. PMID 22006130